CLINICAL TRIAL: NCT03371940
Title: Program ACTIVE II: Behavioral Depression Treatment for Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); West Virginia University (Other); Ohio University (Other); University of Michigan (Other)
Responsible Party: Principal Investigator, Mary de Groot, Associate Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1308973934; R18DK092765 (NIH)
Record Dates: First submitted 2017-12-05; First posted 2017-12-13 (Actual); Results first posted 2024-05-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Type2 Diabetes; Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Study subjects were randomly assigned to one of the four groups: talk therapy, exercise, talk therapy + exercise, or usual care. Separate randomization lists were generated by the study statistician for use by each of the three study sites.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Talk therapy (CBT) (Experimental): Participants randomized the talk therapy arm received 10 weeks of CBT or "talk therapy." The goal of CBT was to provide individuals with skills and concepts that they may use to: 1) manage and reduce depressive symptoms; 2) prevent the onset and severity of future depressive episodes; and 3) generalize these skills to diabetes management.
  CBT interventionists facilitated patient management of depressive symptoms by providing participants with:
  * Education about depression and the cognitive-behavioral therapy model;
  * A safe relationship for participants to explore their symptom patterns and try to new tools to address them;
  * Coaching as participants fully engage emotional and behavioral strategies.
  Interventions: Behavioral: Program ACTIVE CBT
- Exercise (EXER) (Experimental): Participants randomized to the exercise arm were enrolled in a 12-week physical activity intervention designed to increase aerobic physical activity. Participants were asked to complete 100 minutes of aerobic activity in Week 1, 125 minutes in Week 2, and 150 minutes per week of physical activity in Weeks 3-12. In addition, participants received 6 exercise training classes in which safe exercise practices were introduced and practiced, free access to a local exercise facility, use of a pedometer, completion of activity logs each week, and received an exercise workbook that addressed social and motivational aspects of physical activity.
  Interventions: Behavioral: Program ACTIVE Exercise
- Talk therapy + exercise (CBT+EXER) (Experimental): Participants randomized to the combination therapy received both talk therapy and exercise concurrently over a 12-week period as detailed above.
  Interventions: Behavioral: Program ACTIVE
- Usual care (UC) (Placebo Comparator): Participants randomized to usual care received no study intervention.
  Interventions: Behavioral: Usual Care - No intervention

INTERVENTIONS:
Behavioral: Program ACTIVE Exercise — Please see the Exercise arm description above.
  Arms: Exercise (EXER)
Behavioral: Program ACTIVE CBT — Please see the Talk Therapy arm description above.
  Arms: Talk therapy (CBT)
Behavioral: Program ACTIVE — Please see the Talk Therapy + Exercise arm description above.
  Arms: Talk therapy + exercise (CBT+EXER)
Behavioral: Usual Care - No intervention — Please see the Usual Care arm description above.
  Arms: Usual care (UC)

SUMMARY:
Program ACTIVE II is a depression treatment study sponsored by the National Institutes of Health, Indiana University, Ohio University and West Virginia University. The purpose of this study is to test the effectiveness of two forms of treatment for depression for adults with type 2 diabetes: talk therapy (counseling) and exercise. Both of these forms of treatment have been proven to be effective in helping people with depression alone. In this study, the investigators will test to see if both of these approaches may be more effective in helping people live depression-free compared to talk therapy, exercise or usual care alone.

DETAILED DESCRIPTION:
Program ACTIVE II is a study funded by the National Institute of Diabetes and Digestive and Kidney Diseases (R18DK092765) designed to test the combined effectiveness of two behavioral treatments for depression in people with type 2 diabetes: individual counseling (cognitive behavioral therapy; CBT) and exercise. While each of these treatment approaches has been tested individually in people with depression, no study has tested the combination of these approaches for people with major depression and type 2 diabetes. These approaches have the potential to work synergistically as a win-win strategy to improve both T2DM and depression outcomes while extending the reach of formal health care treatment strategies for diabetes.

Two primary study aims will be addressed by Program ACTIVE II: 1) to compare changes in glycemic control across intervention groups to UC at POST and 6- and 12-month follow-up assessments; and 2) to compare changes in MDD outcomes across intervention groups (i.e. CBT, EXER, CBT+EXER) to usual care (UC) following intervention (POST) and 6- and 12-month follow-up assessments.

The primary hypotheses are:

1. Diabetes Outcomes. Based on the investigators' pilot data, mean glycemic control (as measured by HbA1c) is expected to improve .4% in participants in the EXER and CBT+EXER treatment conditions at POST compared to baseline [de Groot et al 2009]. Participants assigned to the CBT+EXER treatment are expected to show the greatest improvement in HbA1c followed by those in the EXER group in comparison to the CBT group. No improvement is expected among those assigned to the UC condition.
2. Depression. Participants in the CBT, EXER and CBT+EXER conditions will show clinically significant improvements in BDI and diagnosis of MDD at POST and 6- and 12-month assessments with the greatest improvements expected among those in CBT+EXER condition. Based on pilot data, a) 66% reduction in the number of people who meet DSM-IV criteria for MDD is expected at POST compared to baseline; b) 86-90% percent of cases with MDD remission at POST are expected to remain remitted at the 6-month follow-up; c) severity of depression, as measured by the BDI-II, will significantly decrease from baseline to POST and baseline to follow-up assessments, after co-varying the effect of gender, number of T2DM complications, and exposure to treatment. It is anticipated that participants in the CBT+EXER condition will show the longest remission rates of depression followed by those in EXER and CBT.

   The secondary hypotheses are:
3. Changes in CVD risk factors in the intervention groups compared to UC over time. Physical activity capacity, as measured by the 6-minute walk test (6MWT), will demonstrate the greatest improvements in the CBT+EXER arm, closely followed by the EXER arm at follow-up assessment compared to baseline. Participants in the CBT and UC arms are not expected to show significant improvements. LDL-C is expected to improve at POST in the EXER and CBT+EXER conditions consistent with pilot data.
4. Cost Effectiveness Analyses. The predicted incidence of complications, particularly coronary heart disease (CHD), will be lower among those who receive CBT+EXER condition compared to the CBT, EXER and UC conditions. Further, the costs of this intensive intervention will be offset by a decrease in complication incidence.

ELIGIBILITY:
Inclusion Criteria:

* able to walk without the use of a cane or walker
* diagnosis of type 2 diabetes for at least one year duration or longer
* major depression lasting two weeks or longer

Exclusion Criteria:

* history of diabetic ketoacidosis (DKA)
* history of continuous insulin therapy since diabetes diagnosis
* stage 2 hypertension as defined by JNC VII
* recent cardiac events (e.g., unstable angina, diagnosed angina, PTCA, any cardiac intervention for CAD or tachydysrhythmias in the past six months)
* laser surgery for proliferative retinopathy in the past six months
* history of stroke, lower limb amputation, asensory peripheral neuropathy, aortic stenosis or other sever valvular heart disease, atrial fibrillation, severe COPD (e.g., basal oxygen), class III or IV heart failure
* active suicidal ideation or history of suicide attempt
* history of bipolar disorder
* history of psychotic disorder
* current substance abuse or dependence disorder
* individuals who report the use of a current antidepressant medication for five weeks or less were excluded or deferred for later screening after the 6 week period
* individual who were receiving psychotherapy from a mental health provider for depression were excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2017-07-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Indiana University, Indianapolis, Indiana
  - Ohio University, Athens, Ohio
  - West Virginia University, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] de Groot M, Shubrook J, Schwartz F, Hornsby WG Jr, Pillay Y, Saha C. Program ACTIVE II: Design and Methods for a Multi-Center Community-Based Depression Treatment for Rural and Urban Adults with Type 2 Diabetes. J Diabetes Res Ther. 2015 Aug;1(2):10.16966/2380-5544.108. doi: 10.16966/2380-5544.108. Epub 2015 Aug 5. PMID 27500279
- [Background] de Groot M, Crick KA, Long M, Saha C, Shubrook JH. Lifetime Duration of Depressive Disorders in Patients With Type 2 Diabetes. Diabetes Care. 2016 Dec;39(12):2174-2181. doi: 10.2337/dc16-1145. Epub 2016 Oct 11. PMID 27729427
- [Result] de Groot M, Shubrook JH, Hornsby WG Jr, Pillay Y, Mather KJ, Fitzpatrick K, Yang Z, Saha C. Program ACTIVE II: Outcomes From a Randomized, Multistate Community-Based Depression Treatment for Rural and Urban Adults With Type 2 Diabetes. Diabetes Care. 2019 Jul;42(7):1185-1193. doi: 10.2337/dc18-2400. Epub 2019 May 21. PMID 31221693
- [Result] Kuo S, Ye W, de Groot M, Saha C, Shubrook JH, Hornsby WG Jr, Pillay Y, Mather KJ, Herman WH. Cost-effectiveness of Community-Based Depression Interventions for Rural and Urban Adults With Type 2 Diabetes: Projections From Program ACTIVE (Adults Coming Together to Increase Vital Exercise) II. Diabetes Care. 2021 Apr;44(4):874-882. doi: 10.2337/dc20-1639. Epub 2021 Feb 19. PMID 33608260
- [Derived] Myers BA, Pillay Y, Guyton Hornsby W Jr, Shubrook J, Saha C, Mather KJ, Fitzpatrick K, de Groot M. Recruitment effort and costs from a multi-center randomized controlled trial for treating depression in type 2 diabetes. Trials. 2019 Nov 6;20(1):621. doi: 10.1186/s13063-019-3712-x. PMID 31694682

RESULTS

PARTICIPANT FLOW:
Groups:
- Talk Therapy (CBT): Participants randomized the talk therapy arm received 10 weeks of CBT or "talk therapy." The goal of CBT was to provide individuals with skills and concepts that they may use to: 1) manage and reduce depressive symptoms; 2) prevent the onset and severity of future depressive episodes; and 3) generalize these skills to diabetes management.
  CBT interventionists facilitated patient management of depressive symptoms by providing participants with:
  * Education about depression and the cognitive-behavioral therapy model;
  * A safe relationship for participants to explore their symptom patterns and try to new tools to address them;
  * Coaching as participants fully engage emotional and behavioral strategies.
  Program ACTIVE CBT: Please see the Talk Therapy arm description above.
- Talk Therapy + Exercise (CBT+EXER): Participants randomized to the combination therapy received both talk therapy and exercise as detailed above.
  Program ACTIVE: Please see the Talk Therapy + Exercise arm description above.
Period: Overall Study
Arm/Group | Talk Therapy (CBT) | Exercise (EXER) | Talk Therapy + Exercise (CBT+EXER) | Usual Care (UC)
Started | 36 | 34 | 34 | 36
Completed | 28 | 33 | 31 | 32
Not Completed | 8 | 1 | 3 | 4
Not completed — Withdrawal by Subject | 8 | 1 | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Talk Therapy (CBT) | Exercise (EXER) | Talk Therapy + Exercise (CBT+EXER) | Usual Care (UC) | Total
Number analyzed (Participants) | 36 | 34 | 34 | 36 | 140
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 36 | 34 | 34 | 36 | 140
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.9 (10.9) | 54.6 (10.7) | 57.1 (10.7) | 54.2 (10.4) | 55.95 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 26 | 28 | 27 | 107
  Male | 10 | 8 | 6 | 9 | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 7 | 8 | 7 | 13 | 35
  White | 27 | 25 | 25 | 22 | 99
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 2 | 1 | 6
Region of Enrollment [Number; unit: participants]
  United States | 36 | 34 | 34 | 36 | 140

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c
Description: Based on our pilot data, mean glycemic control (as measured by HbA1c) is expected to improve .4% in participants in the EXER and CBT + EXER treatment conditions at POST (~3 month) compared to baseline (de Groot et al., 2009).
Time Frame: following completion of intervention (POST; ~3 months)
Population: Discrepancies between numbers randomized to each treatment and numbers analyzed are due to factors such as: rejection of treatment, seeking treatment from health care provider instead, transportation issues, scheduling issues or being lost to follow-up.
Measure: Least Squares Mean (Standard Error); unit: percentage of glycosylated hemoglobin
Arm/Group | Talk Therapy (CBT) | Exercise (EXER) | Talk Therapy + Exercise (CBT+EXER) | Usual Care (UC)
Number analyzed (Participants) | 24 | 30 | 25 | 28
percentage of glycosylated hemoglobin | 0.06 (0.13) | -0.03 (0.13) | -0.17 (0.13) | 0.20 (0.13)

2. Primary Outcome: Change in Depression Status - Beck Depression Inventory
Description: The BDI total score is a sum of 21 items (score range 0 - 63) with higher scores indicating greater depression symptomatology. We calculated change scores from baseline to POST (~3 months). Negative values indicate improvements in depression symptoms. Positive values indicate worsened depression symptoms.
Time Frame: following completion of intervention (POST; ~3 months)
Measure: Least Squares Mean (Standard Error); unit: Change in BDI scores
Arm/Group | Talk Therapy (CBT) | Exercise (EXER) | Talk Therapy + Exercise (CBT+EXER) | Usual Care (UC)
Number analyzed (Participants) | 24 | 30 | 25 | 28
Change in BDI scores | -15.24 (1.95) | -14.11 (1.91) | -18.12 (1.81) | -8.21 (1.88)

3. Primary Outcome: Change in Depression Status - Diagnosis of Major Depressive Disorder
Description: Data presented below is the proportion of participants in each treatment arm that achieved partial or full remission from MDD at POST (~3 months) intervention per the Structured Clinical Interview for the DSM-IV.
Time Frame: following completion of intervention (POST; ~3 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Talk Therapy (CBT) | Exercise (EXER) | Talk Therapy + Exercise (CBT+EXER) | Usual Care (UC)
Number analyzed (Participants) | 24 | 30 | 25 | 28
Participants | 16 | 21 | 17 | 9

4. Secondary Outcome: Physical Activity Capacity as Measured by the 6-minute Walk Test (6MWT)
Description: Physical activity capacity as measured by the 6-minute walk test (6MWT, measured in feel walked)
Time Frame: following completion of intervention (POST; ~3 months)
Measure: Least Squares Mean (Standard Error); unit: change in feet walked
Arm/Group | Talk Therapy (CBT) | Exercise (EXER) | Talk Therapy + Exercise (CBT+EXER) | Usual Care (UC)
Number analyzed (Participants) | 24 | 30 | 25 | 28
change in feet walked | -6.16 (33.03) | 65.60 (32.60) | 0.74 (31.48) | 23.68 (33.26)

ADVERSE EVENTS:
Arm/Group | Talk Therapy (CBT) | Exercise (EXER) | Talk Therapy + Exercise (CBT+EXER) | Usual Care (UC)
All-Cause Mortality (participants affected / at risk) | 0/36 | 1/34 | 0/34 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/34 | 0/34 | 0/36
Other Adverse Events (participants affected / at risk) | 3/36 | 13/34 | 11/34 | 9/36
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Talk Therapy (CBT) (N=36) | Exercise (EXER) (N=34) | Talk Therapy + Exercise (CBT+EXER) (N=34) | Usual Care (UC) (N=36)
Adverse Event - Anticipated (General disorders) | 3 (3) | 12 (12) | 11 (11) | 9 (9) — Adverse events due to injuries sustained during exercise such as falls or due to blood sugar anomalies.
Adverse Event - Unanticipated (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Shortness of breath and rapid heartbeat during exercise. EKG was clear.

LIMITATIONS AND CAVEATS:
Predominantly female/relatively small sample sizes in subgroup analyses-may have limited statistical significance. Larger sample size may reach statistical significance.

Confidence intervals observed in the OR of depression remission in CBT group may indicate limited reliability of this estimate.

Participants may not generalize to all adults with T2DM & MDD.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No